CLINICAL TRIAL: NCT01072110
Title: Confocal Laser Endomicroscopy in Patients With Diarrhea
Brief Title: Confocal Laser Endomicroscopy (CLE) in Patients With Diarrhea
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0001
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Diarrhea
Keywords: Patients with diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with diarrhea undergoing endoscopy: Standard video colonoscope.
  Interventions: Procedure: Colonoscopy
- Group 2: Patients with diarrhea undergoing endoscopy.: Confocal laser endomicroscopy (CLE).
  Interventions: Procedure: Confocal Laser Endomicroscopy

INTERVENTIONS:
Procedure: Colonoscopy — Patients will undergo colonoscopy for evaluation of their symptoms.
  Groups: Group 1: Patients with diarrhea undergoing endoscopy
Procedure: Confocal Laser Endomicroscopy — Patients will undergo CLE during their endoscopy. Findings will be compared to group 1.
  Groups: Group 2: Patients with diarrhea undergoing endoscopy.

SUMMARY:
The main objective of this study is to determine the frequency of different gastrointestinal disorders as the cause of diarrhea in patients at a tertiary referral center using confocal laser endomicroscopy.

DETAILED DESCRIPTION:
Background:

Diarrhea is characterized by frequent, loose, and watery bowel movements. Common causes include various gastrointestinal infections (e.g. clostridium difficile, salmonella), inflammatory bowel disease (ulcerative colitis, Crohn´s disease), drugs (e.g. antibiotics) and malabsorption syndromes (e.g. celiac and Whipple's disease). Confocal laser endomicroscopy (CLE) is rapidly emerging as a valuable tool for gastrointestinal endoscopic imaging, enabling the endoscopist to obtain an "optical biopsy" of the gastrointestinal mucosa during the endoscopic procedure.

Scope:

In patients with diarrhea.

Methods:

Patients were randomized in two groups. Group 1: Patients underwent standard video colonoscopy for the evaluation of their symptoms. Group 2: During the endoscopic procedure CLE will be performed additionally.

Procedure:

The patient underwent colonoscopy. In Group 2 patients´ will receive intravenous fluorescein or topical mucosal staining with acriflavin or cresyl violet during the procedure, followed by in-vivo CLE of the tissue. Confocal images are digitally saved and analyzed afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Impaired renal function (Creatinine > 1.2 mg/dl)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Known allergy to fluorescein, acriflavin or cresyl violet
* Residing in institutions (e.g. prison)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a tertiary referral hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of different gastrointestinal disorders as the cause of diarrhea in patients at a tertiary referral center using confocal laser endomicroscopy. | February 2012

SECONDARY OUTCOMES:
To investigate whether CLE has a higher sensitivity and specificity than standard colonoscopy in the diagnosis of the cause of diarrhea. | February 2012

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, M.D., Ph.D., Principal Investigator — Department of Medicine I, University of Erlangen-Nuremberg
Locations (1):
- Erlangen, Germany